CLINICAL TRIAL: NCT03984474
Title: Institute of Sports Medicine of Peking University Third Hospital, Beijing, China
Brief Title: The Clinical Outcome of Anterior Cruciate Ligament Reconstruction
Acronym: RCACLR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Inner Mongolia People's Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jia-kuo yu, Deputy director of Institute of Sports Medicine of Peking University third hospital, Clinical Professor, Peking University Third Hospital
Other Study IDs: ACLR-YJK
Record Dates: First submitted 2019-04-29; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior Cruciate Ligament Reconstruction; Patient-reported outcome; Meniscus; Cartilage
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single bundle group: Age 13-65 when enrolled. Only include isolated ACL rupture. Excluded revision surgery. Excluded bilateral ACL rupture. Excluded the contralateral ACL tear after surgery.
- Double bundle group: Age 13-65 when enrolled. Only include isolated ACL rupture. Excluded revision surgery. Excluded bilateral ACL rupture. Excluded the contralateral ACL tear after surgery.

SUMMARY:
Retrospective cohort study. The investigators evaluated the early, middle and long term effects of different surgical methods of anterior cruciate ligament reconstruction on knee function.

In the evaluation, the investigators focused on the differences between different age groups, different genders and different basic motor states, the differences between early reconstruction and non-early reconstruction, and the differences in clinical outcomes of different surgical methods.

DETAILED DESCRIPTION:
Age 13-65 included. Only include isolated anterior cruciate ligament(ACL) rupture. Excluded revision surgery. Excluded bilateral ACL rupture. Excluded the contralateral ACL tear after surgery. 40 patients at least in each group.

ELIGIBILITY:
Inclusion Criteria:

diagnosis of isolated anterior cruciate ligament rupture

Exclusion Criteria:

combined other ligament damage combined intraarticular injuries

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the anterior cruciate ligament reconstruction in the Peking University Third Hospital during 1999-2017.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2003-01-14 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee(IKDC) score | Preoperative
  The entire IKDC form, which includes a demographic form, current health assessment form, subjective knee evaluation form, knee history form, surgical documentation form, and knee examination form, may be used as separate forms. The knee history form and surgical documentation form are provided for convenience. All researchers are required to complete the subjective knee evaluation and knee examination form. Instructions for scoring the subjective knee evaluation form and the knee examination form are provided on the back of the forms. Total score 100, ≥75 being considered excellent.
International Knee Documentation Committee(IKDC) score | 2 years after surgery
  The entire IKDC form, which includes a demographic form, current health assessment form, subjective knee evaluation form, knee history form, surgical documentation form, and knee examination form, may be used as separate forms. The knee history form and surgical documentation form are provided for convenience. All researchers are required to complete the subjective knee evaluation and knee examination form. Instructions for scoring the subjective knee evaluation form and the knee examination form are provided on the back of the forms. Total score 100, ≥75 being considered excellent.
International Knee Documentation Committee(IKDC) score | 5-8 years after surgery
  The entire IKDC form, which includes a demographic form, current health assessment form, subjective knee evaluation form, knee history form, surgical documentation form, and knee examination form, may be used as separate forms. The knee history form and surgical documentation form are provided for convenience. All researchers are required to complete the subjective knee evaluation and knee examination form. Instructions for scoring the subjective knee evaluation form and the knee examination form are provided on the back of the forms. Total score 100, ≥75 being considered excellent.
International Knee Documentation Committee(IKDC) score | 10-15 years after surgery
  The entire IKDC form, which includes a demographic form, current health assessment form, subjective knee evaluation form, knee history form, surgical documentation form, and knee examination form, may be used as separate forms. The knee history form and surgical documentation form are provided for convenience. All researchers are required to complete the subjective knee evaluation and knee examination form. Instructions for scoring the subjective knee evaluation form and the knee examination form are provided on the back of the forms. Total score 100, ≥75 being considered excellent.
International Knee Documentation Committee(IKDC) score | an average of 20 year
  The entire IKDC form, which includes a demographic form, current health assessment form, subjective knee evaluation form, knee history form, surgical documentation form, and knee examination form, may be used as separate forms. The knee history form and surgical documentation form are provided for convenience. All researchers are required to complete the subjective knee evaluation and knee examination form. Instructions for scoring the subjective knee evaluation form and the knee examination form are provided on the back of the forms. Total score 100, ≥75 being considered excellent.
KT-2000 test | 2 years after surgery
  It is a kind of joint measuring instrument used to determine the anteroposterior stability of knee joint. The contrast between the uninjured side and the surgical measurement showed that the difference of ≤3mm was considered excellent.
KT-2000 test | 5-8 years after surgery
  It is a kind of joint measuring instrument used to determine the anteroposterior stability of knee joint. The contrast between the uninjured side and the surgical measurement showed that the difference of ≤3mm was considered excellent.
KT-2000 test | 10-15 years after surgery
  It is a kind of joint measuring instrument used to determine the anteroposterior stability of knee joint. The contrast between the uninjured side and the surgical measurement showed that the difference of ≤3mm was considered excellent.
KT-2000 test | an average of 20 year
  It is a kind of joint measuring instrument used to determine the anteroposterior stability of knee joint. The contrast between the uninjured side and the surgical measurement showed that the difference of ≤3mm was considered excellent.
Magnatic Resonance Imaging evaluation | Preoperative
  All patients undergoing anterior cruciate ligament reconstruction underwent MRI imaging evaluation of both knees. Use International Cartilage Repair Society(ICRS) score to evaluate, total score is 12, classified into four grades,grade Ⅰ: normal (12), grade Ⅱ: nearly normal (8-11), grade Ⅲ: abnormal (4-7), grade Ⅳ: severely abnormal (1-3).
Magnatic Resonance Imaging evaluation | 2 years after surgery
  All patients undergoing anterior cruciate ligament reconstruction underwent MRI imaging evaluation of both knees. Use International Cartilage Repair Society(ICRS) score to evaluate, total score is 12, classified into four grades,grade Ⅰ: normal (12), grade Ⅱ: nearly normal (8-11), grade Ⅲ: abnormal (4-7), grade Ⅳ: severely abnormal (1-3).
Magnatic Resonance Imaging evaluation | 5-8 years after surgery
  All patients undergoing anterior cruciate ligament reconstruction underwent MRI imaging evaluation of both knees. Use International Cartilage Repair Society(ICRS) score to evaluate, total score is 12, classified into four grades,grade Ⅰ: normal (12), grade Ⅱ: nearly normal (8-11), grade Ⅲ: abnormal (4-7), grade Ⅳ: severely abnormal (1-3).
Magnatic Resonance Imaging evaluation | 10-15 years after surgery
  All patients undergoing anterior cruciate ligament reconstruction underwent MRI imaging evaluation of both knees. Use International Cartilage Repair Society(ICRS) score to evaluate, total score is 12, classified into four grades,grade Ⅰ: normal (12), grade Ⅱ: nearly normal (8-11), grade Ⅲ: abnormal (4-7), grade Ⅳ: severely abnormal (1-3).
Magnatic Resonance Imaging evaluation | an average of 20 year
  All patients undergoing anterior cruciate ligament reconstruction underwent MRI imaging evaluation of both knees. Use International Cartilage Repair Society(ICRS) score to evaluate, total score is 12, classified into four grades,grade Ⅰ: normal (12), grade Ⅱ: nearly normal (8-11), grade Ⅲ: abnormal (4-7), grade Ⅳ: severely abnormal (1-3).

SECONDARY OUTCOMES:
Skeletal force line and various angles by X-ray evaluation | Preoperative
  X-ray was used to evaluate the skeletal force line and various angles of patients. Use Qvadriceps Angle to evaluate quadriceps force line and patellar ligament force line. The normal Angle is 18-22° for the adult standing position.Above or below this range is considered abnormal.
Skeletal force line and various angles by X-ray evaluation | 2 years after surgery
  X-ray was used to evaluate the skeletal force line and various angles of patients. Use Qvadriceps Angle to evaluate quadriceps force line and patellar ligament force line. The normal Angle is 18-22° for the adult standing position.Above or below this range is considered abnormal.
Skeletal force line and various angles by X-ray evaluation | 5-8 years after surgery
  X-ray was used to evaluate the skeletal force line and various angles of patients. Use Qvadriceps Angle to evaluate quadriceps force line and patellar ligament force line. The normal Angle is 18-22° for the adult standing position.Above or below this range is considered abnormal.
Skeletal force line and various angles by X-ray evaluation | 10-15 years after surgery
  X-ray was used to evaluate the skeletal force line and various angles of patients. Use Qvadriceps Angle to evaluate quadriceps force line and patellar ligament force line. The normal Angle is 18-22° for the adult standing position.Above or below this range is considered abnormal.
Skeletal force line and various angles by X-ray evaluation | an average of 20 year
  X-ray was used to evaluate the skeletal force line and various angles of patients. Use Qvadriceps Angle to evaluate quadriceps force line and patellar ligament force line. The normal Angle is 18-22° for the adult standing position.Above or below this range is considered abnormal.

OTHER OUTCOMES:
Biomechanical analysis of human gait | 2 years after surgery
  Biomechanical analysis of human gait was performed in all patients under load and no load conditions. Step length, cadence, speed and Angle of patients were evaluated, and then the assessment reports were summarized into "similar" or "abnormal" ones with normal people.
Biomechanical analysis of human gait | 5-8 years after surgery
  Biomechanical analysis of human gait was performed in all patients under load and no load conditions. Step length, cadence, speed and Angle of patients were evaluated, and then the assessment reports were summarized into "similar" or "abnormal" ones with normal people.
Biomechanical analysis of human gait | 10-15 years after surgery
  Biomechanical analysis of human gait was performed in all patients under load and no load conditions. Step length, cadence, speed and Angle of patients were evaluated, and then the assessment reports were summarized into "similar" or "abnormal" ones with normal people.
Biomechanical analysis of human gait | an average of 20 year
  Biomechanical analysis of human gait was performed in all patients under load and no load conditions. Step length, cadence, speed and Angle of patients were evaluated, and then the assessment reports were summarized into "similar" or "abnormal" ones with normal people.
Rotational torque of knee by Biodex system isokinetic testing | 2 years after surgery
  Use Biodex system(BIODEXMEDICALSYSTEMS,INC) to assess the increase or decrease in the amount of rotational torque applied to the patient's limb velocity as it accelerates and decelerates. The equal-velocity quadriceps moment of the operating leg up to 85% of the uninjured side is considered normal.
Rotational torque of knee by Biodex system isokinetic testing | 5-8 years after surgery
  Use Biodex system(BIODEXMEDICALSYSTEMS,INC) to assess the increase or decrease in the amount of rotational torque applied to the patient's limb velocity as it accelerates and decelerates. The equal-velocity quadriceps moment of the operating leg up to 85% of the uninjured side is considered normal.
Rotational torque of knee by Biodex system isokinetic testing | 10-15 years after surgery
  Use Biodex system(BIODEXMEDICALSYSTEMS,INC) to assess the increase or decrease in the amount of rotational torque applied to the patient's limb velocity as it accelerates and decelerates. The equal-velocity quadriceps moment of the operating leg up to 85% of the uninjured side is considered normal.
Rotational torque of knee by Biodex system isokinetic testing | an average of 20 year
  Use Biodex system(BIODEXMEDICALSYSTEMS,INC) to assess the increase or decrease in the amount of rotational torque applied to the patient's limb velocity as it accelerates and decelerates. The equal-velocity quadriceps moment of the operating leg up to 85% of the uninjured side is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kuo Yu, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Mao Z, Wang J, Wang Y, Jiang D, Wang X, Wang H, Lin L, Liu Y, Zeng L, Yu J. Double-bundle anterior cruciate ligament reconstruction technique has advantages in chondroprotection and knee laxity control compared with single-bundle technique : A long-term follow-up with a minimum of 12 years. Knee Surg Sports Traumatol Arthrosc. 2021 Sep;29(9):3105-3114. doi: 10.1007/s00167-020-06350-5. Epub 2020 Nov 20. PMID 33216188